CLINICAL TRIAL: NCT07344194
Title: Dual-Site Transcranial Magnetic Stimulation of the Supplementary Motor Area and Cerebellum for the Treatment of Essential Tremor
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: São Paulo State University (Other)
Responsible Party: Principal Investigator, ANANDA CAROLINA MORAES DE FALCONE, Principal Investigator, São Paulo State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 81190724.8.0000.0068
Record Dates: First submitted 2026-01-07; First posted 2026-01-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Essential Tremor
Keywords: essential tremor; rTMS; movement disorders; non-invasive neuromodulation
MeSH Terms: conditions — Essential Tremor; Movement Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The intervention is active rTMS stimulation (1 Hz, 110% of resting motor threshold) over the supplementary motor area in 24 trains with 3-second inter-train intervals, followed by high-frequency stimulation of the cerebellar cortex (10 Hz, 90% of resting motor threshold) delivered in 12 trains with 3-second inter-train intervals
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization will be performed by an independent researcher not involved in treatment delivery or outcome assessment. The randomization assignment will be communicated only to the investigator responsible for administering the transcranial magnetic stimulation (TMS).
  Clinical evaluations will be conducted by a separate investigator who is blinded to treatment allocation.
  Participants in the control group will receive sham stimulation using a sham coil positioned over the same scalp location as the active stimulation. The sham coil does not produce a magnetic field but is combined with a secondary coil placed near the participant to generate auditory stimulation, reproducing the sound characteristics of active TMS. Stimulation parameters and session duration will be identical to those used in the active group, in order to maintain participant blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-site rTMS over SMA (1 Hz, 110% RMT) and cerebellum (10 Hz, 90% RMT) for 5 days. (Experimental): Sham stimulation over SMA and cerebellum using inactive coil with sound simulation for 5 days.
  Interventions: Device: Dual-site repetitive transcranial magnetic stimulation (rTMS) of the supplementary motor area and cerebellum
- Sham (Sham Comparator): The sham intervention replicates the anatomical targeting, sequence, session duration, and acoustic characteristics of the active dual-site rTMS protocol without delivering an effective magnetic field. An inactive coil is positioned over the same supplementary motor area and cerebellar targets, while sound simulation is used to mimic active stimulation, ensuring maintenance of blinding and comparability with the active intervention.
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Dual-site repetitive transcranial magnetic stimulation (rTMS) of the supplementary motor area and cerebellum — This intervention consists of a sequential dual-site repetitive transcranial magnetic stimulation (rTMS) protocol targeting two interconnected nodes of the tremor network. Low-frequency stimulation (1 Hz) is first applied over the supplementary motor area at 110% of the resting motor threshold to modulate cortical motor drive, followed by high-frequency stimulation (10 Hz) over the cerebellar cortex at 90% of the resting motor threshold to modulate abnormal cerebellar output. Stimulation is delivered over five consecutive daily sessions using standardized anatomical localization and identical session duration across participants.
  Sham Intervention
  The sham intervention replicates the anatomical targeting, sequence, session duration, and acoustic characteristics of the active dual-site rTMS protocol without delivering an effective magnetic field. An inactive coil is positioned over the same supplementary motor area and cerebellar cortex
  Arms: Dual-site rTMS over SMA (1 Hz, 110% RMT) and cerebellum (10 Hz, 90% RMT) for 5 days.
Device: Transcranial Magnetic Stimulation Sham — The sham intervention replicates the anatomical targeting, sequence, session duration, and acoustic characteristics of the active dual-site rTMS protocol without delivering an effective magnetic field. An inactive coil is positioned over the same supplementary motor area and cerebellar targets, while sound simulation is used to mimic active stimulation, ensuring maintenance of blinding and comparability with the active intervention.
  Other Names: Sham
  Arms: Sham

SUMMARY:
Essential tremor is a common movement disorder that causes involuntary shaking, mainly during voluntary actions such as writing or holding objects. Recent research suggests that essential tremor is not caused by a single brain area, but by abnormal activity within a network that includes the cerebellum and motor areas of the brain. However, most non-invasive brain stimulation studies to date have targeted only one brain region and have shown inconsistent clinical benefits.

This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the effects of a dual-site transcranial magnetic stimulation (rTMS) protocol targeting the supplementary motor area (SMA) and the cerebellum in patients with essential tremor that does not respond adequately to standard medications. The study is based on previous pilot data showing meaningful tremor reduction using combined stimulation of these two brain regions.

Participants will receive five sessions of rTMS, consisting of low-frequency stimulation over the SMA followed by high-frequency stimulation over the cerebellum. The main hypothesis is that this combined approach will lead to an immediate and sustained improvement in action tremor of the dominant upper limb, measured up to four weeks after treatment. Secondary outcomes include quality of life, safety, side effects, and changes in brain excitability associated with tremor improvement.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, parallel-group phase II clinical trial designed to investigate the effects of dual-site repetitive transcranial magnetic stimulation (rTMS) in patients with medication-refractory essential tremor. The trial is conducted at the University of São Paulo.

Participants are randomized to receive either active or sham stimulation over five consecutive daily sessions. The active intervention consists of sequential stimulation of two interconnected nodes of the tremor network. Low-frequency rTMS (1 Hz, 110% of resting motor threshold) is first applied over the supplementary motor area in 24 trains with 3-second inter-train intervals, followed by high-frequency stimulation of the cerebellar cortex (10 Hz, 90% of resting motor threshold) delivered in 12 trains with 3-second inter-train intervals. The protocol is designed to modulate cortical motor drive and cerebellar output within the cerebello-thalamo-cortical circuit.

The stimulation parameters and dual-site approach were selected based on neurophysiological and neuroimaging evidence supporting a network-based model of essential tremor, as well as on pilot data demonstrating clinically meaningful tremor reduction following combined stimulation of the supplementary motor area and cerebellum.

Participants are evaluated at baseline, immediately after completion of the stimulation protocol, and during follow-up to assess clinical effects, safety, and neurophysiological changes associated with the intervention. This study aims to further characterize the therapeutic potential of network-targeted rTMS in essential tremor and to inform future neuromodulation strategies in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, aged 18 to 80 years; women of childbearing potential must not be pregnant.
* Diagnosis of Essential Tremor with a score greater than 2 on items 5 or 6 of the Fahn-Tolosa-Marin Tremor Rating Scale despite optimized medical therapy.
* Medication-refractory tremor, defined as prior use of both first-line medications (propranolol and primidone) at maximally tolerated doses without adequate tremor control.
* Ability to provide written informed consent in accordance with institutional policies.
* Ability to comply with all study procedures and follow-up assessments as defined by the study protocol.

Exclusion Criteria:

* Unstable or untreated psychiatric disorders.
* Inability to provide informed consent.
* Uncontrolled medical conditions, including but not limited to uncontrolled diabetes mellitus, hypertension, symptomatic pulmonary disease, or symptomatic cardiac disease.
* Concomitant participation in another investigational drug or device study.
* Pregnancy or breastfeeding.
* Presence of an implanted deep brain stimulation (DBS) system.
* History of epilepsy not adequately controlled, defined as seizure-free for less than 5 years.
* Presence of a cardiac pacemaker.
* Presence of metallic implants in any part of the body that are contraindicated for rTMS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in Action Tremor Severity of the Dominant Upper Limb | baseline (pre-stimulation), at the end of the stimulation protocol, 4 weeks after the last session
  Assessed using items 5 and 6 of the Fahn-Tolosa-Marin Tremor Rating Scale, evaluated by a blinded examiner.

CONTACTS AND LOCATIONS:
Locations (1):
- Sao Paulo University, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in publications will be made available upon reasonable request to the corresponding author, following publication. Data sharing will be subject to approval by the institutional ethics committee and execution of a data use agreement, in accordance with applicable data protection regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 2 years after the publication of results
Access Criteria: Requests for access to de-identified individual participant data will be considered for scientifically sound research purposes that are consistent with the objectives of the original study. Proposed analyses must not conflict with participant consent or institutional ethical approvals. Requests should include a brief research proposal outlining the study objectives, planned analyses, and statistical methods.
  All requests will be reviewed by the study investigators and, when required, by the institutional ethics committee. Data sharing will be contingent upon approval of the proposed analyses and execution of a data use agreement in accordance with institutional policies and applicable data protection regulations. Approved data will be shared in a de-identified format through secure data transfer methods.